CLINICAL TRIAL: NCT02469961
Title: Dexmedetomidine vs Propofol TIVA and Interscalene Block for Shoulder Surgeries in a Beach Chair Sitting Position
Brief Title: Dexmedetomidine vs Propofol TIVA (Total Intravenous Anesthesia) and Interscalene Block
Acronym: TIVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Piyush Gupta, MD, Clinical Director, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10/07/VA07
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2016-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): Participants will receive an interscalene block and be sedated with dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Other: Interscalene block
- Propofol (Active Comparator): Participants will receive an interscalene block and be sedated with propofol
  Interventions: Drug: Propofol; Other: Interscalene block

INTERVENTIONS:
Drug: Dexmedetomidine — Participants will receive an interscalene block and will be sedated with Dexmedetomidine and compared to sedation with propofol
  Other Names: precedex
  Arms: dexmedetomidine
Drug: Propofol — Participants will receive an interscalene block and be sedated with Propofol and compared to sedation with Dexmedetomidine
  Other Names: diprivan
  Arms: Propofol
Other: Interscalene block — Interscalene block is used for the main anesthetic for the case

SUMMARY:
The standard hospital procedure calls for the patient to undergo Interscalene block under ultrasound with or without nerve stimulation guidance prior to going to operating room (OR). The block utilizes a 40 ml mixture of 0.5% Ropivacaine and Lidocaine 1.5%. At this time the patient receives preliminary sedation with Midazolam 1mg IV and Fentanyl 50 mcg IV. The participant is then brought to the OR and prolonged sedation is initiated, randomly using either Dexmedetomidine or Propofol.

The primary objective of the present study is to use Dexmedetomidine for sedation, and compare the outcomes with Propofol sedation. The investigators will enroll 50 patients for this study.

Our hypothesis is that Dexmedetomidine will cause fewer episodes of intermittent apnea, and reduced need for supplemental medication for sedation, compared to Propofol

DETAILED DESCRIPTION:
The anesthesia provided during shoulder surgery commonly uses a combination of regional and intravenous (IV) anesthetic medications. The current drug of choice for IV sedation is Propofol. Although. it is a good anesthetic, incidence of intermittent apnea makes the use of it problematic in cases where the head of the patient is less accessible to the anesthesiologist, as is in sitting beach char position. Dexmedetomidine is a FDA approved drug, which has a very stable cardiovascular and respiratory profile. It has been successfully used for Neurological and Vascular cases and in Intensive care units. The primary objective of the present study is to use Dexmedetomidine for sedation, and compare the outcomes with Propofol sedation. The investigators' will enroll 50 patients for this study. Using a computer program the participants will be randomized into two equal groups to receive either Dexmedetomidine or Propofol.

The standard hospital procedure calls for the patient to undergo Interscalene block under ultrasound with or without nerve stimulation guidance prior to going to operating room (OR). The block utilizes a 40 ml mixture of 0.5% Ropivacaine and Lidocaine 1.5%. At this time the patient receives preliminary sedation with Midazolam 1mg IV and Fentanyl 50 mcg IV. The participant is then brought to the OR and prolonged sedation is initiated, randomly using either Dexmedetomidine or Propofol.

Dexmedetomidine infusion is initiated with a bolus of 1 mcg/kg is given over 10 min as patient is being positioned, and the sedation is maintained with Dexmedetomidine at 0.7- 1.0 mcg/kg/hr during the surgery. Propofol infusion is started at 100mcg/kg/min, and maintained with Propofol at 50-120mcg/kg/min, during the surgery.

In each group the investigators will record the incidence of respiratory depression/hypoxia, hemodynamic stability, frequency of airway manipulation, cardiovascular effects, need for anesthetic supplementation of Dexmedetomidine, post anesthesia care unit (PACU) discharge time, the need for postoperative pain medication, post operative complications, like nausea/vomiting.

Significant differences between the two groups will be evaluated using unpaired t-test for numerical variables, and Chi-square test or Z test for categorical variables.

The investigators hypothesis is that Dexmedetomidine will cause fewer episodes of intermittent apnea, and reduced need for supplemental medication for sedation, compared to Propofol

ELIGIBILITY:
Inclusion Criteria:

Participants scheduled for shoulder arthroscopies in the beach chair sitting position.

Participants who received a successful interscalene block.

Exclusion Criteria:

Failed interscalene block. Refusal to participate in the study. Allergy to the study drugs. Participants that need a secure airway.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: piyush Gupta, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Mehta PP, Kochhar G, Kalra S, Maurer W, Tetzlaff J, Singh G, Lopez R, Sanaka MR, Vargo JJ. Can a validated sleep apnea scoring system predict cardiopulmonary events using propofol sedation for routine EGD or colonoscopy? A prospective cohort study. Gastrointest Endosc. 2014 Mar;79(3):436-44. doi: 10.1016/j.gie.2013.09.022. Epub 2013 Nov 9. PMID 24219821
- [Result] Venn RM, Hell J, Grounds RM. Respiratory effects of dexmedetomidine in the surgical patient requiring intensive care. Crit Care. 2000;4(5):302-8. doi: 10.1186/cc712. Epub 2000 Jul 31. PMID 11056756

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidne: Participants will receive an interscalene block and be sedated with dexmedetomidine
  Dexmedetomidine: Participants will receive an interscalene block and will be sedated with Dexmedetomidine and compared to sedation with propofol
  Interscalene block: Interscalene block is used for the main anesthetic for the case
- Propofol: Participants will receive an interscalene block and be sedated with propofol
  Propofol: Participants will receive an interscalene block and be sedated with Propofol and compared to sedation with Dexmedetomidme
  Interscalene block: Interscalene block is used for the main anesthetic for the case
Period: Overall Study
Arm/Group | Dexmedetomidne | Propofol
Started | 25 | 25
Completed | 21 | 24
Not Completed | 4 | 1
Not completed — Physician Decision | 4 | 1

BASELINE CHARACTERISTICS:
Population: 45
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Propofol | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Need an Airway Intervention.
Description: airway manipulation or repositioning: apnea, oral airway, adjust head
Time Frame: Participants will be followed from the start of sedation until discharge: approximately 3-5 hr
Measure: Number; unit: participants
Groups:
- Dexmedetomidine: Number of patients required airway manipulation
- Propofol: Number of patients required airway manipulations
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 21 | 24
participants | 0 | 5

2. Secondary Outcome: Post Anesthesia Care Unit (PACU) Length of Stay
Description: length of stay in minutes in the Post Anesthesia Care Unit before discharge
Time Frame: Arrival in the PACU until discharge either to home or to a hospital in-patient bed approximately 1-3 hr after the operation
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 21 | 24
Minutes | 159 (12) | 126 (12)

3. Secondary Outcome: Number of Participants That Have Either Bradycardia or Hypotension
Description: Number of participants observed with Bradycardia or Hypotension who required intervention
Time Frame: Participants will be followed from the start of sedation until discharge: approximately 3-5 hr
Population: Number of patients who had Bradycardia or hypotension
Measure: Number; unit: participants
Groups:
- Propofol: Patients who received Propofol
- Dexmedetomidine: Patients who received Dexmedetomidine
Arm/Group | Propofol | Dexmedetomidine
Number analyzed (Participants) | 24 | 21
participants | 4 | 5

4. Secondary Outcome: Total Narcotic Used by Each Participant
Description: the use for morphine and/or fentanyl and or Demerol converted to morphine equivalents
Time Frame: Participants will be followed from the start of sedation until discharge: approximately 3-5 hr
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | Dexmedetomidine | Propofol
Number analyzed (Participants) | 21 | 24
Microgram | 7.1 (23.9) | 9 (24.2)

ADVERSE EVENTS:
Time Frame: Study was conducted for one year and four months
Arm/Group | Dexmedetomidine | Propofol
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

LIMITATIONS AND CAVEATS:
There was no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No